CLINICAL TRIAL: NCT05977569
Title: Physiological and Sensory Responses to Prolonged Fasting in Humans
Acronym: PRO-FAST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Bath (Other)
Collaborators: University of Nottingham (Other)
Responsible Party: Principal Investigator, James Betts, Professor, University of Bath
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PF
Record Dates: First submitted 2021-09-07; First posted 2023-08-04 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-07

CONDITIONS: Fasting; Metabolic Disturbance; Energy Supply; Deficiency; Adiposity
MeSH Terms: conditions — Fasting; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prolonged Fasting (Experimental): All participants are asked to act as their own control prior to being asked to undergo 3 days of fasting.
  Interventions: Other: Prolonged Fasting

INTERVENTIONS:
Other: Prolonged Fasting — Participants are asked to refrain from caloric intake for 3 days following a period of habitual lifestyle assessment and metabolic assessment.

SUMMARY:
This study aims to establish the metabolic/molecular response in both adipose tissue and skeletal muscle as well as sensory experiences (pain, fatigue, drive) to prolonged fasting of 3 days duration. Participants will undergo sequential meal assessment before and after a 3 day fast with measures taken throughout each fasting day.

DETAILED DESCRIPTION:
This study will employ a single-arm, non-randomised design in which participants will act as their own control prior to undergoing 3 days of fasting. The control phase includes 3 days of habitual energy balance assessment before coming into the laboratory for baseline meal testing with blood, muscle, and adipose samples as well as anthropometric assessment.

Participants will then be provided with a standardised lunch to be consumed around midday and a standardised dinner to be consumed at 2000 h.

Participants will then be asked to refrain from caloric intake for 3 days until they return to the laboratory for follow up measures.

Participants will be provided with monitoring equipment throughout the 3 days of fasting and will be asked to provide a blood sample at 0800 h each day alongside self recording of blood pressure, weight, and urinary ketones each day. On the middle day (day 2) participants will also be asked to come into the lab to provide a blood sample at 2000 h.

The follow up visit will be identical to that performed before the fast, including meal testing, blood, muscle, and adipose samples.

ELIGIBILITY:
Inclusion Criteria:

* • Body mass index 20.0-29.9 kg∙m-2

  * Age 18-45 years
  * Willing to abstain from food intake for just over 3 days (~82 hours)
  * Able and willing to provide informed consent and safely comply with study procedures
  * Females to maintain record of regular menstrual cycle phase or contraceptive use
  * No anticipated changes in lifestyle during the study (e.g. holidays or exercise programmes)

Exclusion Criteria:

* • Any reported condition or behaviour deemed either to pose undue personal risk to the participant or introduce bias

  * Any diagnosed metabolic disease (e.g. type 1 or type 2 diabetes)
  * Any reported use of substances which may pose undue personal risk to the participants or introduce bias into the experiment
  * Pregnancy
  * Breastfeeding
  * Lifestyle not conforming to standard sleep-wake cycle (e.g. shift worker)
  * History of eating disorders (e.g. anorexia)
  * Any reported recent (<6 months) change in body mass (± 3%)
  * Uncontrolled hyperthyroidism
  * Advanced cerebrovascular insufficiency or dementia
  * Advanced liver or kidney insufficiency
  * History of migraine and or headache
  * Psychotic disorders
  * Unstable or severe coronary artery disease
  * Retinal detachment
  * Duodenal or stomach ulcer
  * Cancer and malignant disease
  * Regular use of Non-steroidal anti-inflammatory drugs (NSAIDs)
  * Use of Systemic corticoids
  * Use of Antihypertensives (especially beta-blockers and diuretics)
  * Use of Antidiabetics
  * Use of Anti-coagulants
  * Use of Psychotropics (especially neuroleptics and lithium)
  * Use of Anticonvulsants.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Estimated)
Dates: Start 2021-06-28 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Change in postprandial insulin responses | 3 days
  Change in postprandial insulin (mmol/L) response to a standardised meal before and after 3 days of fasting.

SECONDARY OUTCOMES:
Change in circulating glycerol and non-esterified fatty acids | 1 day, 2 days, 3 days
  Change in indices of lipolysis from adipose tissue in response to prolonged fasting (Glycerol mmol/L; NEFA mmol/L)
Change in Autophagy | 3 days
  Change in autophagic flux in response to prolonged fasting, assessed in skeletal muscle and circulating neutrophils.
Change in plasma lactate | 1 day, 2 days, 3 days
  Change in plasma lactate in response to prolonged fasting (indices of Cori cycle)
Change in plasma pyruvate | 1 day, 2 days, 3 days
  Change in plasma pyruvate in response to prolonged fasting (indices of Cori cycle)
Change in ketosis. | 1 day, 2 days, 3 days.
  Change in urinary (acetoacetate) ketones in response to prolonged fasting.
Change in ketosis. | 1 day, 2 days, 3 days.
  Change in circulating (beta-hydroxybutyrate) ketones in response to prolonged fasting.
Change in body mass | 1 day, 2 days, 3 days.
  Change in body mass, pre-post, and during the prolonged fast.
Change in blood pressure | 1 day, 2 days, 3 days.
  Change in blood pressure pre-, post-, and during the prolonged fast
Change in interstitial fluid glucose concentrations | 1 day, 2 days, 3 days.
  Change in interstitial fluid glucose concentrations pre-, post-, and during the prolonged fast (assessed via continual glucose monitoring)
Change in amino acid metabolism | 3 days.
  Change in amino acid metabolism (i.e. BCAAs and ketoacids) in skeletal muscle
Change in amino acid metabolism | 3 days.
  Change in amino acid metabolism (i.e. BCAAs and ketoacids) in adipose tissue
Change in amino acid metabolism | 3 days.
  Change in amino acid metabolism (i.e. BCAAs and ketoacids) in circulation
Change in postprandial glucose responses. | 3 days.
  Change in postprandial glucose (mmol/L) response to a standardised meal before and after 3 days of fasting.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bath, Bath, Somerset, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-09-23): https://cdn.clinicaltrials.gov/large-docs/69/NCT05977569/Prot_SAP_000.pdf
  • Informed Consent Form (2020-11-23): https://cdn.clinicaltrials.gov/large-docs/69/NCT05977569/ICF_001.pdf